CLINICAL TRIAL: NCT00631111
Title: Ibuprofen 400 mg Effervescent Tablet Dental Pain Study II
Brief Title: Study Evaluating the Efficacy of an Ibuprofen Effervescent Tablet in the Treatment of Post-Surgical Dental Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AI-07-02
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2009-08-10 (Estimated); Status verified 2009-07

CONDITIONS: Pain
Keywords: dental pain; analgesic; NSAID; ibuprofen; aspirin
MeSH Terms: conditions — Pain; Toothache | interventions — Ascorbic Acid; Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: effervescent ibuprofen tablets
- 2 (Active Comparator)
  Interventions: Drug: effervescent Aspirin plus Vitamin C tablets
- 3 (Active Comparator)
  Interventions: Drug: ibuprofen tablets
- 4 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: effervescent ibuprofen tablets
  Arms: 1
Drug: effervescent Aspirin plus Vitamin C tablets
  Arms: 2
Drug: ibuprofen tablets
  Arms: 3
Drug: placebo
  Arms: 4

SUMMARY:
Evaluation of the efficacy and safety of a single dose of an ibuprofen effervescent tablet in the treatment of pain following third molar extraction in comparison to single doses of placebo, standard ibuprofen tablets, and effervescent aspirin plus vitamin C tablets.

ELIGIBILITY:
Inclusion:

* Moderate or severe post-operative pain following surgical extraction of two or more third molars, at least one of which must be a partial or complete bony mandibular impaction
* In general good health with no contraindications to the study medication or rescue medication (tramadol or acetaminophen + hydrocodone)
* Use of only short-acting local anesthetics with or without vasocontrictor and/or nitrous oxide

Exclusion:

* Presence of a serious medical condition (e.g., poorly controlled hypertension, diabetes, or hyper-/hypo-thyroidism; significantly impaired renal, cardiac, or hepatic function)
* Acute localized dental alveolar infection at the time of surgery that could confound the post-surgical evaluation
* Females who are pregnant, lactating, of child-bearing potential, or post-menopausal for less than 2 years and not using a medically-approved method of contraception

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 270 (Actual)
Dates: Start 2007-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Sum of pain relief and pain intensity difference scores | 8 hours

SECONDARY OUTCOMES:
Time to meaningful pain relief | 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Austin, Texas, United States